CLINICAL TRIAL: NCT06638099
Title: Increasing Use of Continuous Glucose Monitors Among Patients With Type 2 Diabetes
Brief Title: Increasing CGM Use Among Patients With T2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HS-2024-0026; UH3MD018353 (NIH)
Record Dates: First submitted 2024-10-05; First posted 2024-10-15 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Diabetes; Diabetes Mellitus; Diabetes Mellitus Type 2; Diabetes Mellitus Type 2 (T2DM)
Keywords: Diabetes Mellitus Type 2; Continuous Glucose Monitor; FQHC Intervention; health care providers; CGM Education
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthcare Prescribers Exposed to CGM Prescriber Toolkit Training (Experimental): Participants in this arm will include qualified healthcare prescribers (MDs, DOs, PAs, NPs, etc.) and staff who treat patients with Type 2 diabetes in primary care settings who will receive in depth training using a study-developed prescriber toolkit. The toolkit covers important information including current clinical practice guidelines, eligibility criteria, provider documentation requirements and scripts for discussing CGM use with their patient population. The impact of the training will be evaluated by examining changes in CGM prescription rates for patients with Type 2 diabetes seen in primary care before and after the training is delivered. Secondarily, Participants will be surveyed pre- and post-training to elicit prescribing knowledge and attitudes towards CGM use.
  Interventions: Behavioral: CGM Toolkit Prescriber Training
- Healthcare Prescribers Not Exposed to CGM Prescriber Toolkit Training (No Intervention): Participants in this arm are prescribers (MDs, DOs, PAs, NPs, etc.) and staff who will NOT receive in depth training using a study-developed prescriber toolkit.

INTERVENTIONS:
Behavioral: CGM Toolkit Prescriber Training — A CGM prescription toolkit was created for prescribing clinicians and staff that includes written guidance on CGM eligibility criteria, instructions for screening patients for eligibility using EHR records and during healthcare visits, recommended provider documentation templates to address all required eligibility criteria for insurance coverage of CGM device and supplies (e.g., Medicare, Medicaid), sample scripts for communicating with patients about the purpose and use of CGM, and patient-level frequently asked questions (FAQs), including free resources available to learn more about CGM benefits, where/how to acquire CGM, and determining out-of-pocket costs. The toolkit will be introduced during a 20 minute initial training session and reinforced during a 10 minute booster training approximately one month after initial training
  Arms: Healthcare Prescribers Exposed to CGM Prescriber Toolkit Training

SUMMARY:
Study Overview:

This interventional study aims to assess whether training healthcare professionals (HCPs) increases the number of continuous glucose monitor (CGM) prescriptions for patients with Type 2 Diabetes in a Federally Qualified Health Center serving a predominantly Hispanic/Latino population.

Research Questions:

Does HCP training enhance CGM prescription rates in a primary care setting? Does receiving a CGM prescription lead to improved Type 2 Diabetes control, as measured by Hemoglobin A1c levels? What barriers do patients face when prescribed and using CGMs? Given the significant impact of CGMs on diabetes management, this project seeks to improve CGM utilization among eligible patients through a focused intervention for HCPs and evaluate diabetes outcomes for those who do and do not receive a CGM.

Methodology:

HCPs and staff from three clinics within the same healthcare system will undergo a brief, in-person training on current clinical guidelines and insurance eligibility for CGMs. A booster session will follow about one month later to reinforce learning and address any prescribing challenges.

Training efficacy will be evaluated by comparing CGM prescription rates before and after training using electronic health records. HCPs will complete pre- and post-training surveys to assess changes in knowledge, beliefs, and prescribing practices related to CGMs. Additionally, a small subset of prescribers will participate in interviews about their experiences with CGM prescriptions four months post-training.

Patient Recruitment and Surveys:

Patients with Type 2 Diabetes will be recruited for surveys at baseline, and at 3 and 6 months. These surveys will gather information on their diabetes management experience, levels of diabetes distress, and whether CGM discussions occurred with their primary care provider. Participants who received CGM prescriptions will share their experiences and any barriers encountered. A subset will also be invited for interviews to further explore their CGM experiences.

Conclusion:

This study seeks to fill a crucial gap in understanding how HCP training influences CGM prescription rates and the associated diabetes management outcomes, ultimately aiming to enhance diabetes care for a vulnerable population.

DETAILED DESCRIPTION:
Background & Significance: Approximately 30 million adults in the U.S. suffer from diabetes, a chronic condition with serious long-term health and social consequences. Diabetes is a leading cause of death and disability across the country that disproportionately burdens minoritized ethnoracial, low-income, and rural populations-such as in the border-area region of Imperial County, CA where diabetes rates far exceed state and national averages.Continuous glucose monitoring (CGM) is increasingly recognized as a valuable tool for patients with Type 1 and Type 2 Diabetes (T1D and T2D, respectively), with use of the technology associated with improved disease management, reduced diabetes distress, and healthcare costs. Unfortunately, while clinical practice guidelines recommend use of CGM in diabetes care, inequities in CGM use threaten to exacerbate existing diabetes disparities. For instance, patients from minoritized ethnoracial groups, particularly Hispanic and Black patients, are less likely to use CGM than non-Hispanic white patients.

Disparities in CGM use may be attributed to a variety of factors; However, the most common barrier reported by both patients and providers is limited uptake due to perceived cost. Research has shown that providers may not prescribe CGM due to concerns about costs and their lack of knowledge about insurance eligibility requirements. Fortunately, recent expansions in insurance coverage mean costs may no longer prohibit access to CGM for low-income patients who meet clinical eligibility criteria. Notwithstanding, many providers may not prescribe CGM even to those who qualify for coverage. This may be particularly true among primary care providers who increasingly serve as the primary point of care for patients with diabetes living in rural and medically underserved areas without access to an endocrinologist. A study of over 600 HCPs showed that only 38.6% had ever prescribed CGM, but nearly two-thirds said they would be likely to do so with increased education on CGM or consultation on insurance requirements. Thus, educating HCP on current CGM clinical practice recommendations and insurance coverage eligibility requirements could greatly improve CGM prescriptions in clinics serving low-income and ethnoracially diverse patients.

While increasing CGM prescriptions is an important step to providing more equitable access to CGM, additional intervention may be needed to ensure patients from historically marginalized communities can access and use the devices. More specifically, once prescribed, CGM effectiveness is contingent on patients' acquiring, applying and using the device. Research has shown that patients may share their providers' uncertainty over coverage eligibility requirements and out-of-pocket costs associated with CGM use; a study of over 1,500 patients with T1D found the most reported concerns about using CGM were insurance coverage and costs. If not addressed, cost concerns could impede patients from acquiring CGMs even if prescribed by their healthcare provider (HCP).

Given the potential impact of CGM on diabetes management, efforts to increase CGM uptake are critically needed, especially in historically marginalized and under-resourced regions without access to diabetes specialty care. Strategies such as educating HCP on current CGM eligibility criteria and insurance costs and improving patient education on costs may be effective in increasing initial CGM uptake and ultimately improving patient outcomes. However, no prior studies have evaluated the impact of these strategies in low-resource, primary care settings, or with Hispanic/Latino patients. Existing studies have also primarily focused on CGM use and impact in patients with T1D rather than T2D. The proposed project will fill this gap by evaluating the impact of a system-level, provider-focused intervention on CGM prescription rates and diabetes outcomes for eligible patients with T2D of a large Federally-Qualified Health Center in Imperial County, California.

The project will be guided by the following aims:

1.Determine whether the proportion of T2D patients who are prescribed CGM significantly increases following a system-level CGM intervention that is implemented sequentially in three different clinics. HCPs and staff will participate in a training and receive a CGM prescription toolkit, including procedures for determining clinical eligibility, insurance documentation templates, scripts for communication with patients, and patient education materials with information about CGM benefits, how and where to acquire the device, and any anticipated out-of-pocket costs. CGM prescription rates will be extracted from electronic health records (EHR) to determine changes over time. H1: CGM prescription rate for T2D patients will increase significantly after the intervention.

1a: Evaluate impact of toolkit training on knowledge and attitudes towards CGM among HCP/Staff. H2: Knowledge and attitudes towards CGM will significantly improve following completion of the toolkit training.

2. Compare changes in A1C values over time between T2D patients who do and do not receive a CGM. A1C values will be extracted from the EHR to compare changes over time among patients with T2D who received and filled a new CGM prescription vs. never received or did not fill their prescription. H0: Patients who use CGM will show significantly greater improvement in A1C values over 6 months compared to those who did not use CGM.

2a. Determine whether the impact of CGM use on A1C is mediated by changes in diabetes distress. H2: Reductions in diabetes distress will mediate the relationship between CGM use and A1C among patients.

3.Identify factors that influence CGM uptake among healthcare providers, staff, and patients. Providers, staff, and patients will complete interviews about their experiences with CGM post-intervention. H3: NA.

Research Design & Methods:

The study aims will be achieved in a three-phase, three-year project. This study will be conducted in collaboration with Innercare, which is a federally-qualified health center in Imperial County, CA, and participants will include healthcare professionals (HCPsl including prescribing clinicians and their staff) and patients recruited from the three largest Innercare clinics in Imperial County: Brawley, El Centro, Calexico. In Phase 1, the investigators will evaluate a systems-level intervention (CGM prescription toolkit and associated training for HCPs and staff) designed to improve CGM prescription rates among patients with T2D in primary care clinics (Aim 1, 1a, 3). In Phase 2, the impact of CGM use on diabetes management among patients with T2D will be evaluated through an examination of A1C laboratory values extracted from the electronic health records (EHR) of patients who were prescribed and received a CGM during the study period (Aim 2). Additionally, the mechanisms of action for CGM will be explored by examining diabetes distress as a mediator between CGM use and A1C values among a subset of patients who complete a self-report survey that will be linked to their EHR data (Aim 2a). In Phase 3, patients will participate in one-on-one interviews about their experiences with CGM, including challenges and facilitators to accessing and using the technology (Aim 3).

ELIGIBILITY:
Participant Eligibility:

Inclusion:

* adults 18 years or older,
* have been diagnosed with T2D at least one year prior to recruitment,
* are a current patient of one of the three participating Innercare Clinics with no -
* plans to discontinue their care at Innercare within the next 6 months,
* can understand and speak in English or Spanish,
* have telephone access,
* do not plan to move out of the area within the next 6 months.

Exclusion:

* Plans to move out of the area in the next 6 months
* Patients with newly diagnose diabetes mellitus (less than one year), diabetes insipidus, diabetes type 1 or gestational diabetes.

Provider/Staff Eligibility:

Inclusion

* 18 years or older,
* able to read and write in English,
* currently employed at one of the participating Innercare clinics (Brawley, El Centro, Calexico),
* currently be treating at least one adult patient for T2D, scheduled to complete the CGM toolkit training. Exclusion
* Personnel without experience providing care to adult patients with T2D in primary care settings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
CGM prescription rates | From training until month 6
  Determine if the proportion of patients with T2D who are prescribed CGM increases following the intervention as compared to pre-intervention data

SECONDARY OUTCOMES:
HCP/Staff Knowledge and Attitudes Towards CGM Use & Prescribing Behavior in Target Population | Pre-training to Month 3
  Use of repeated measures survey assessment of HCP/staff knowledge, attitudes, and prescribing behaviors towards CGM use in target population. Survey includes 16 measures assessing HCP/staff knowledge of different diabetes management metrics, attitudes towards CGM, and prescribing behaviors. Knowledge is assessed using three measures that assess current glucose management practices for adult patients with Type 1 or Type 2 diabetes and awareness of different diabetes metrics. Attitudes towards CGM are assessed using a 6-item Likert measure, with values ranging from 1-4, and higher scores indicating more positive attitudes towards CGM. HCP/staff CGM prescribing behaviors are assessed using four measures that address whether providers currently prescribe CGM for patients (yes/no), criteria evaluated prior to prescribing CGM (open-ended), and strategies for introducing CGMs to patients or addressing patient questions about CGM (check all that apply).
Effect of CGM Prescription on HgbA1C | Receipt of CGM Prescription to Month 6
  Measure impact of CGM use on diabetes management among patients with T2D through examination of A1C laboratory values extracted from the electronic health records (EHR) of patients who were prescribed and received a CGM during the study period. HgbA1c will be extracted for individuals who have received a CGM prescription from their PCP. A baseline HgbA1C value will be recorded for the patient within 3 months prior to the prescription and then 3- 6 months following the prescription.
Effect of CGM on Individual Diabetes Distress Among Patients with T2D | Receipt of CGM Prescription to month 6
  Evaluate mechanisms of action of CGM on diabetes distress as a mediator between CGM use and A1C values among a subset of patients who complete a self-report survey that will be linked to their EHR data. Diabetes distress: The 17-item Diabetes Distress Scale is a widely used tool for assessing diabetes distress and has been validated in both English and Spanish. Participants report the frequency they experience 17 symptoms in the past 7 such as, "Feeling that diabetes is taking up too much of my mental and physical energy every day." All items from this scale are averaged to create a mean scale score.
Challenges and Facilitators to CGM Uptake in Patients with T2D | Receipt of CGM to Month 6
  Determine challenges and facilitators to accessing and using CGM technology in patients with T2D through one-to-one telephone interviews aimed at collecting qualitative data regarding experiences with CGM. Specifically, patients who were prescribed, acquired, and used a CGM will be asked to describe their experiences discussing CGM with their provider and with obtaining and using the CGM; patients who received but did not fill a CGM prescription will be asked to elucidate reasons for non-use; and patients that never received a CGM prescription will be asked about their knowledge and attitudes towards CGM and factors that might affect use.

OTHER OUTCOMES:
Participant Experience with Prescribing, Acquiring and/or Using a CGM. | Clinic Implementation to Month 9
  In one-on-one telephone interviews lasting 20-30 minutes, patients will be asked to discuss their various experiences with CGM. Specifically, patients who were prescribed, acquired, and used a CGM will be asked to describe their experiences discussing CGM with their provider and with obtaining and using the CGM; patients who received but did not fill a CGM prescription will be asked to elucidate reasons for non-use; and patients that never received a CGM prescription will be asked about their knowledge and attitudes towards CGM and factors that might affect use.
HCP/Staff Experiences with Prescribing & Monitoring CGM use in Target Population | Toolkit Training to Month 6
  In one-on-one telephone interviews lasting 20-30 minutes, patients will be asked to discuss their various experiences with CGM. Specifically, HCP/Staff experience with prescribing and facilitating access to CGM for target population.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Schmied,, PhD, Principal Investigator — San Diego State University; Shiloh Williams, PhD RN, Principal Investigator — San Diego State University
Locations (2):
- United States (2):
  - Innercare Inc, El Centro, California
  - Innercare, Inc, El Centro, California

IPD SHARING:
Plan to Share IPD: Yes
Undecided
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: To be determined
Access Criteria: To be determined

REFERENCES:
- [Background] Ni K, Tampe CA, Sol K, Richardson DB, Pereira RI. Effect of CGM Access Expansion on Uptake Among Patients on Medicaid With Diabetes. Diabetes Care. 2023 Feb 1;46(2):391-398. doi: 10.2337/dc22-1287. PMID 36480729
- [Background] Vrany EA, Hill-Briggs F, Ephraim PL, Myers AK, Garnica P, Fitzpatrick SL. Continuous glucose monitors and virtual care in high-risk, racial and ethnic minority populations: Toward promoting health equity. Front Endocrinol (Lausanne). 2023 Jan 25;14:1083145. doi: 10.3389/fendo.2023.1083145. eCollection 2023. PMID 36761197
- [Background] Davidson JA. The increasing role of primary care physicians in caring for patients with type 2 diabetes mellitus. Mayo Clin Proc. 2010 Dec;85(12 Suppl):S3-4. doi: 10.4065/mcp.2010.0466. Epub 2010 Nov 24. No abstract available. PMID 21106869
- [Background] Tanenbaum ML, Adams RN, Hanes SJ, Barley RC, Miller KM, Mulvaney SA, Hood KK. Optimal Use of Diabetes Devices: Clinician Perspectives on Barriers and Adherence to Device Use. J Diabetes Sci Technol. 2017 May;11(3):484-492. doi: 10.1177/1932296816688010. Epub 2017 Jan 10. PMID 28745093
- [Background] Lanning MS, Tanenbaum ML, Wong JJ, Hood KK. Barriers to Continuous Glucose Monitoring in People With Type 1 Diabetes: Clinician Perspectives. Diabetes Spectr. 2020 Nov;33(4):324-330. doi: 10.2337/ds19-0039. PMID 33223770
- [Background] Tanenbaum ML, Hanes SJ, Miller KM, Naranjo D, Bensen R, Hood KK. Diabetes Device Use in Adults With Type 1 Diabetes: Barriers to Uptake and Potential Intervention Targets. Diabetes Care. 2017 Feb;40(2):181-187. doi: 10.2337/dc16-1536. Epub 2016 Nov 29. PMID 27899489
- [Background] Walker AF, Hood KK, Gurka MJ, Filipp SL, Anez-Zabala C, Cuttriss N, Haller MJ, Roque X, Naranjo D, Aulisio G, Addala A, Konopack J, Westen S, Yabut K, Mercado E, Look S, Fitzgerald B, Maizel J, Maahs DM. Barriers to Technology Use and Endocrinology Care for Underserved Communities With Type 1 Diabetes. Diabetes Care. 2021 Jul;44(7):1480-1490. doi: 10.2337/dc20-2753. Epub 2021 May 17. PMID 34001535
- [Background] Smith MB, Albanese-O'Neill A, Macieira TGR, Yao Y, Abbatematteo JM, Lyon D, Wilkie DJ, Haller MJ, Keenan GM. Human Factors Associated with Continuous Glucose Monitor Use in Patients with Diabetes: A Systematic Review. Diabetes Technol Ther. 2019 Oct;21(10):589-601. doi: 10.1089/dia.2019.0136. Epub 2019 Aug 20. PMID 31335196
- [Background] Warman M, Fillippi M, Manning B, Oser T, Nease D, Hall T, Oser S, Carroll J. Continuous glucose monitoring for primary care patients with diabetes: Barriers, facilitators, & resources to support access. Ann Fam Med. 2022 Apr 1;20(20 Suppl 1):2689. doi: 10.1370/afm.20.s1.2689. PMID 36857171
- [Background] Oser TK, Hall TL, Dickinson LM, Callen E, Carroll JK, Nease DE Jr, Michaels L, Oser SM. Continuous Glucose Monitoring in Primary Care: Understanding and Supporting Clinicians' Use to Enhance Diabetes Care. Ann Fam Med. 2022 Nov-Dec;20(6):541-547. doi: 10.1370/afm.2876. PMID 36443083
- [Background] Kanbour S, Jones M, Abusamaan MS, Nass C, Everett E, Wolf RM, Sidhaye A, Mathioudakis N. Racial Disparities in Access and Use of Diabetes Technology Among Adult Patients With Type 1 Diabetes in a U.S. Academic Medical Center. Diabetes Care. 2023 Jan 1;46(1):56-64. doi: 10.2337/dc22-1055. PMID 36378855
- [Background] Isaacs D, Bellini NJ, Biba U, Cai A, Close KL. Health Care Disparities in Use of Continuous Glucose Monitoring. Diabetes Technol Ther. 2021 Sep;23(S3):S81-S87. doi: 10.1089/dia.2021.0268. PMID 34546086
- [Background] Fantasia KL, Wirunsawanya K, Lee C, Rizo I. Racial Disparities in Diabetes Technology Use and Outcomes in Type 1 Diabetes in a Safety-Net Hospital. J Diabetes Sci Technol. 2021 Sep;15(5):1010-1017. doi: 10.1177/1932296821995810. Epub 2021 Mar 10. PMID 33719610
- [Background] Aljedaani SM, Siddiqui AS, Raja-Khan N. 678-P: Racial and Ethnic Disparities in CGM Use among Adults with Diabetes. Diabetes. 2022;71(Supplement_1).
- [Background] Blonde L, Umpierrez GE, Reddy SS, McGill JB, Berga SL, Bush M, Chandrasekaran S, DeFronzo RA, Einhorn D, Galindo RJ, Gardner TW, Garg R, Garvey WT, Hirsch IB, Hurley DL, Izuora K, Kosiborod M, Olson D, Patel SB, Pop-Busui R, Sadhu AR, Samson SL, Stec C, Tamborlane WV Jr, Tuttle KR, Twining C, Vella A, Vellanki P, Weber SL. American Association of Clinical Endocrinology Clinical Practice Guideline: Developing a Diabetes Mellitus Comprehensive Care Plan-2022 Update. Endocr Pract. 2022 Oct;28(10):923-1049. doi: 10.1016/j.eprac.2022.08.002. Epub 2022 Aug 11. PMID 35963508
- [Background] Polonsky WH, Hessler D, Ruedy KJ, Beck RW; DIAMOND Study Group. The Impact of Continuous Glucose Monitoring on Markers of Quality of Life in Adults With Type 1 Diabetes: Further Findings From the DIAMOND Randomized Clinical Trial. Diabetes Care. 2017 Jun;40(6):736-741. doi: 10.2337/dc17-0133. Epub 2017 Apr 7. PMID 28389582
- [Background] Norman GJ, Paudel ML, Parkin CG, Bancroft T, Lynch PM. Association Between Real-Time Continuous Glucose Monitor Use and Diabetes-Related Medical Costs for Patients with Type 2 Diabetes. Diabetes Technol Ther. 2022 Jul;24(7):520-524. doi: 10.1089/dia.2021.0525. Epub 2022 Apr 27. PMID 35230158
- [Background] Karter AJ, Parker MM, Moffet HH, Gilliam LK, Dlott R. Association of Real-time Continuous Glucose Monitoring With Glycemic Control and Acute Metabolic Events Among Patients With Insulin-Treated Diabetes. JAMA. 2021 Jun 8;325(22):2273-2284. doi: 10.1001/jama.2021.6530. PMID 34077502
- [Background] Ida S, Kaneko R, Murata K. Utility of Real-Time and Retrospective Continuous Glucose Monitoring in Patients with Type 2 Diabetes Mellitus: A Meta-Analysis of Randomized Controlled Trials. J Diabetes Res. 2019 Jan 15;2019:4684815. doi: 10.1155/2019/4684815. eCollection 2019. PMID 30775385
- [Background] Gavin JR, Bailey CJ. Real-World Studies Support Use of Continuous Glucose Monitoring in Type 1 and Type 2 Diabetes Independently of Treatment Regimen. Diabetes Technol Ther. 2021 Sep;23(S3):S19-S27. doi: 10.1089/dia.2021.0211. PMID 34165343
- [Background] Beck RW, Bergenstal RM. Continuous Glucose Monitoring for Type 2 Diabetes: How Does It Compare with Type 1 Diabetes? Diabetes Technol Ther. 2022 Mar;24(3):153-156. doi: 10.1089/dia.2021.0374. Epub 2021 Oct 13. No abstract available. PMID 34569811
- [Background] California Department of Public Health. 2017-2018 Border Health Status Report to the Legislature: Diabetes. 2019.
- [Background] Bullard KM, Cowie CC, Lessem SE, Saydah SH, Menke A, Geiss LS, Orchard TJ, Rolka DB, Imperatore G. Prevalence of Diagnosed Diabetes in Adults by Diabetes Type - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Mar 30;67(12):359-361. doi: 10.15585/mmwr.mm6712a2. PMID 29596402

DOCUMENTS (1):
  • Informed Consent Form (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT06638099/ICF_000.pdf